CLINICAL TRIAL: NCT02042911
Title: A Multicenter, Open-label Phase II Study of SyB L-0501 in Patients With Chronic Lymphocytic Lymphoma
Brief Title: Efficacy and Safety Study of SyB L-0501 for Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012003
Record Dates: First submitted 2013-12-17; First posted 2014-01-23 (Estimated); Results first posted 2016-03-29 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

ARMS (1):
- SyB L-0501 (Experimental)
  Interventions: Drug: SyB L-0501

INTERVENTIONS:
Drug: SyB L-0501 — SyB L-0501 is administered at 100 mg/m2/day by intravenous infusion on Day 1 and Day 2 followed by 26 days of monitoring. This is considered to be one cycle and may be repeated up to 6 cycles. Dose administration can be delayed or discontinued from the second cycle as necessary according to adverse events and the results of monitoring during the previous cycle, but dose reduction is permitted from the 3rd cycle.

SUMMARY:
The purpose of this study is to investigate safety and efficacy of SyB L-0501 after 2-day intravenous infusion at a dose of 100 mg/m2/day to patients with chronic lymphocytic leukemia.

ELIGIBILITY:
Inclusion Criteria

Patients meeting all of the following criteria are to be included in the study:

1. Patients aged between 20 and 80 years (at the time of registration)
2. Patients who have provided written consent in person for participation in this study
3. Patients with Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 2
4. Patients who are expected to survive for at least 3 months
5. Patients who are naive to or not suitable for fludarabine therapy
6. Patients who are documented with chronic lymphocytic leukemia on the basis of International Workshop on Chronic Lymphocytic Leukaemia guideline (IWCLL) guideline:

   * The presence of ≥ 5000/mm3 monoclonal mature B-lymphocytes in the peripheral blood
   * ≤ 55 % atypical lymphocytes, prolymphocyte-like cells, and lymphoblasts with prominent nucleoli
   * For monoclonal mature B-lymphocytes, at least one of the B-cell specific differentiation antigens (Cluster of differentiation (CD) 19, CD 20, and CD 23) and CD 5 is positive by flow cytometry
7. Patients in Stage C or stage B with active disease based on Binet staging system (at the time of registration)

   * Decision to start treatment should be made upon IWCLL guideline criteria.
   * Active disease is defined to meet at least one of the following criteria.

     1. Progression and/or worsening of anemia and/or thrombocytopenia caused by decreased bone marrow function.
     2. Massive (6 cm below the left costal margin) or progressive or symptomatic splenomegaly
     3. Massive nodes (≥10 cm in longest diameter) or progressive or symptomatic lymphadenopathy
     4. Progressive lymphocytosis with an increase of > 50% over a 2-month period, or lymphocyte doubling time of less than 6 months
     5. Autoimmune anemia and/or thrombocytopenia poorly responsive to corticosteroids or other standard therapy
     6. B symptoms Weight loss > 10% within the previous 6 months Fevers of greater than 38.0° C for 2 or more weeks without other evidence of infection Night sweats
8. Patients with 2 or less regimens of previous chemotherapy including antibody therapy. Corticosteroid monotherapy is not counted.
9. Patients with adequately maintained organ functions (e.g., bone marrow, heart, lung, liver, and kidney functions)

   * Neutrophil count: ≥ 1,000 /mm3
   * Aspartate aminotransferase(AST) Glutamic oxaloacetic transaminase(GOT): ≤ 3.0 times the upper limit of normal range at each site
   * Alanine aminotransferase (ALT) Glutamic pyruvic transaminase(GPT): ≤ 3.0 times the upper limit of normal range at each site
   * Total bilirubin: ≤ 1.5 times the upper limit of normal range at each site
   * Serum creatinine: ≤ 1.5 times the upper limit of normal range at each site
   * Partial pressure of O2 (PaO2): ≥ 65 mmHg
   * No abnormalities which require treatment are detected on ECG
   * Left ventricular ejection fraction (LVEF) (echocardiography): ≥ 55%

Exclusion Criteria:

Patients who fall under any one of the following criteria are to be excluded

1. Patients who have been without treatment for less than 4 weeks after prior treatment. For patients treated with antibody therapy or underwent hematopoietic stem cell transplantation, for 3 months after prior treatment
2. Patients who enrolled other clinical studies within 4 weeks before registration for this study
3. Patients who received allogeneic stem cell transplantation in the past
4. Patients with defective p53 (17p-) confirmed by chromosome analysis (Fluorescence in situ hybridization (Fish) method)
5. Patients who are clinically diagnosed with Richter's syndrome
6. Patients with infiltration to the central nervous system (CNS) or patients with clinical symptoms of suspected infiltration to the CNS
7. Patients with multiple primary cancers or patients with a history of other malignant tumors within past 5 years, except for basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix or gastrointestinal tract
8. Patients with serious bleeding tendencies (e.g., disseminated intravascular coagulation (DIC))
9. Patients with, or confirmed in the past to have had, interstitial lung disease or pulmonary fibrosis
10. Patients with, or confirmed in the past to have had, autoimmune hemolytic anemia responds to corticosteroid therapy
11. Patients with any of the following complications

    * serious cardiac disease (e.g., myocardial infarction, ischemic heart disease, or arrhythmia requiring treatment)
    * serious, active infections (requiring intravenous administration of antibiotics, antifungal drugs, or antiviral drugs)
    * hepatic or renal dysfunction
    * accumulation of pleural effusion, pericardial effusion, or peritoneal effusion
    * uncontrollable serious gastrointestinal disease, endocrine disorder, or mental illness
12. Patients who received SyB L-0501 in the past
13. Patients with allergies to mannitol
14. Patients who need cytokine preparations such as erythropoietin or granulocyte colony stimulating factor (G-CSF) or blood transfusions at registration for this study
15. Patients positive for HIV antibody or Hepatitis C virus (HCV) antibody
16. Patients positive for Hepatitis B surface (HBs) antigen. Patients with negative results will also be checked for Hepatitis B core (HBc) antibody and HBs antibody. If either of the test results is positive, measure Hepatitis B virus (HBV)-DNA and exclude the patients with results above sensitivity
17. Patients with clinical symptom of cytomegalovirus (CMV) infection, except asymptomatic patients with CMV positive
18. Patients who are pregnant, who may possibly be pregnant, or lactating
19. Patients who do not agree to practice contraception. Male: During investigational product administration and until 6 months after final administration Female: During investigational product administration and until 4 months after final administration
20. Patients with drug addiction, narcotics addiction, and/or alcohol dependency
21. Patients otherwise judged by the investigator or sub-investigator to be unsuitable for inclusion in this study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toshihiko Nagase, Study Director — SymBio Pharmaceuticals
Locations (6):
- Japan (6):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Fukuyama, Hiroshima
  - Research Site, Kagoshima, Kagoshima-ken
  - Research Site, Isehara, Kanagawa
  - Research Site, Izumo, Shimane
  - Research Site, Minato-ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- SyB L-0501: SyB L-0501: SyB L-0501 is administered at 100 mg/m^2/day by intravenous infusion on Day 1 and Day 2 followed by 26 days of monitoring. This is considered to be one cycle and may be repeated up to 6 cycles. Dose administration can be delayed or discontinued from the second cycle as necessary according to adverse events and the results of monitoring during the previous cycle, but dose reduction is permitted from the 3rd cycle.
Period: Overall Study
Arm/Group | SyB L-0501
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | SyB L-0501
Number analyzed (Participants) | 10
Age, Customized [Number; unit: participants]
  <65 years | 2
  >=65 years | 8
Gender [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Prior therapy [Number; unit: participants]
  Absent | 8
  Present | 2
ECOG performance status [Number; unit: participants] — The criteria of Eastern Cooperative Oncology Group (ECOG) performance status are shown as below:
  0: Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  participants
    0 | 8
    1 | 2
    2 | 0
Clinical disease stage (Binet Staging System) [Number; unit: participants] — The criteria of clinical disease stage (Binet Staging System) are shown as below:
  Stage A: Hb ≧ 10g/dL + platelet count ≧ 100,000 /mm3 and fewer than 2 areas of enlarged lymphoid tissue Stage B: Hb ≧ 10g/dL + platelet count ≧ 100,000 /mm3 and 3 or more areas of enlarged lymphoid tissue
  Stage C: Hb < 10g/dL and/or platelet count < 100,000 /mm3 :
  Area of lymphoid tissue (one side in the case of two sides) includes: 1) head and neck; 2) axilla; 3) groin; 4) spleen and 5) liver.
  participants
    A | 0
    B | 3
    C | 7
Medical history [Number; unit: participants]
  Absent | 4
  Present | 6
Complication [Number; unit: participants] — Pathological processes or events developing in the course of a primary disease or condition.
  participants
    Absent | 1
    Present | 9
Fluorescence in situ hybridization (FISH) detection of trisomy 12 [Number; unit: participants]
  Absent | 8
  Present | 2
FISH detection of del (13q14) [Number; unit: participants]
  Absent | 5
  Present | 5
FISH detection of del (11q22-23) [Number; unit: participants]
  Absent | 10
  Present | 0
FISH detection of del (17p13) [Number; unit: participants]
  Absent | 10
  Present | 0
FISH detection of immunoglobulin heavy chain (IgH)/CyclinD1 (CCND1) (BCL1) t (11; 14) [Number; unit: participants]
  Absent | 10
  Present | 0
Somatic hypermutation (SHM) analysis of immunoglobulin heavy chain variable (IgVH) genes [Number; unit: participants]
  Absent | 1
  Present | 9
Diagnosis of chronic lymphocytic leukemia (CLL) [Number; unit: participants]
  Yes | 10
  No | 0
Lymphadenopathy [Number; unit: participants]
  Absent | 2
  Present | 8
Hepatomegaly [Number; unit: participants]
  Absent | 5
  Present | 5
Splenomegaly [Number; unit: participants]
  Absent | 1
  Present | 9
B symptoms (Weight Loss) [Number; unit: participants] — >10% weight loss in the last 6 month
  participants
    Absent | 10
    Present | 0
B symptoms (Fever) [Number; unit: participants] — Persistent or recurrent fever of unknown origin > 38 °C for 2 weeks or more
  participants
    Absent | 10
    Present | 0
B symptoms (Night Sweats) [Number; unit: participants]
  Absent | 8
  Present | 2
Presence of cluster of differentiation (CD) 5 antigen [Number; unit: participants] — Presence of CD5 antigen (positive or negative) was evaluated by flow cytometry in the diagnosis of CLL.
  participants
    Negative (-) | 0
    Positive (+) | 10
Presence of CD19 antigen [Number; unit: participants] — Presence of CD19 antigen (positive or negative) was evaluated by flow cytometry in the diagnosis of CLL.
  participants
    Negative (-) | 0
    Positive (+) | 10
Presence of CD20 antigen [Number; unit: participants] — Presence of CD20 antigen (positive or negative) was evaluated by flow cytometry in the diagnosis of CLL.
  participants
    Negative (-) | 0
    Positive (+) | 10
Presence of CD23 antigen [Number; unit: participants] — Presence of CD23 antigen (positive or negative) was evaluated by flow cytometry in the diagnosis of CLL.
  participants
    Negative (-) | 2
    Positive (+) | 8
Presence of Igκ [Number; unit: participants] — Presence of Igκ (positive or negative) was evaluated by flow cytometry in the diagnosis of CLL.
  participants
    Negative (-) | 4
    Positive (+) | 6
Presence of Igλ [Number; unit: participants] — Presence of Igλ (positive or negative) was evaluated by flow cytometry in the diagnosis of CLL.
  participants
    Negative (-) | 6
    Positive (+) | 4
Marrow examination for lymphoid nodules [Number; unit: participants] — Bone marrow aspirate and biopsy was done for assessment of response to evaluate ³30% of the nucleated cells being lymphocyte in the bone marrow sample.
  participants
    Absent | 5
    Present | 5
Marrow examination for infiltration [Number; unit: participants] — Bone marrow aspirate and biopsy was done for assessment of response to evaluate the focal infiltration in the bone marrow sample.
  participants
    Absent | 1
    Present | 9
Height [Mean (Standard Deviation); unit: cm] | 162.03 (5.03)
Body weight [Mean (Standard Deviation); unit: kg] | 56.51 (9.43)
Body surface area [Mean (Standard Deviation); unit: m^2] | 1.592 (0.134)
Age [Mean (Standard Deviation); unit: years] | 69.8 (8.9)

OUTCOME MEASURES:

1. Primary Outcome: Response Rate [Complete Remission (CR) +Complete Remission / Incomplete (CRi) + Nodular Partial Remission (nPR) + Partial Remission (PR)] Based on International Workshop on Chronic Lymphocytic Leukemia (IWCLL) Guideline
Description: The criteria for CR, CRi, nPR and PR based on IWCLL guideline are shown below. For the criteria for nPR and PR, please refer to the description of NCI-WG response rate (CR+nPR+PR).
  CR: Assessment should be made at least 8 weeks after completion of administration.
  1. Absence of significant lymphadenopathy (lymph nodes greater than 1.5 cm in diameter)
  2. No hepatomegaly or splenomegaly
  3. Absence of B symptoms
  4. Meet the following laboratory test values;
     * lymphocyte count in peripheral blood: <4.0×10^9/L
     * neutrophil count: >1.5×10^9/L
     * platelet count: 100×10^9/L
     * hemoglobin: 11.0 g/dL without transfusions
  5. less than 30% of nucleated cells are lymphocytes (confirmed by bone marrow aspiration and no lymphoid nodules).
  6. No new lesion emergence
  CRi: Fulfills all of the following criteria
  * Delayed anemia, thrombocytopenia, or neutropenia is observed.
  * Fulfills all CR criteria other than 4).
  * Delayed symptoms are all judged to be caused by drug.
Time Frame: Up to 30 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SyB L-0501
Number analyzed (Participants) | 10
Percentage of participants | 60.0 [26.2 to 87.8]

2. Secondary Outcome: National Cancer Institute-sponsored Working Group (NCI-WG) Response Rate (CR+nPR+PR) Based on IWCLL Guideline
Description: The criteria for nPR and PR based on IWCLL guideline are shown below.
  nPR: Fulfills all CR criteria other than residual lymphoid nodules confirmed by bone marrow examination.
  PR: Fulfills two or more items from Group A and one or more items from Group B for a minimal duration of 8 weeks.
  Group A;
  1. 50% or greater reduction in lymphocyte count in peripheral blood from baseline
  2. 50% or greater reduction (size reduction) in Sum of the products of the greatest diameters (SPD) and no new lesion emergence or no new enlarged lymph node
  3. A decrease in the size of the liver and/or spleen by 50% more
  4. A decrease in marrow infiltration or lymphoid nodules by 50% more Group B;
  1) Neutrophil count >1.5×10^9/L or 50% improvement from baseline 2) Platelet count >100×10^9/L or 50% improvement from baseline 3) Hemoglobin 11.0 g/dL or 50% improvement from baseline without transfusions
Time Frame: Up to 30 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SyB L-0501
Number analyzed (Participants) | 10
Percentage of participants | 60.0 [26.2 to 87.8]

3. Secondary Outcome: Complete Remission Rate (CR+CRi) Based on IWCLL Guideline
Time Frame: Up to 30 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SyB L-0501
Number analyzed (Participants) | 10
Percentage of participants | 20.0 [2.5 to 55.6]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: The period from the first day of the study drug administration (Day1) to progressive disease (PD), recurrence/relapse, or death.
Time Frame: Up to 30 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SyB L-0501
Number analyzed (Participants) | 10
months | NA [NA to NA] — Because no events were reported at the time of analysis for PFS.

5. Secondary Outcome: Duration of Remission
Description: The period from the day of CR or PR confirmation to recurrence/relapse.
Time Frame: Up to 30 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SyB L-0501
Number analyzed (Participants) | 10
months | NA [NA to NA] — Because no events were reported at the time of analysis for the duration of remission.

6. Secondary Outcome: Overall Survival (OS)
Description: The period from the date of patient registration to the date of death.
Time Frame: Up to 30 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SyB L-0501
Number analyzed (Participants) | 10
months | NA [NA to NA] — Because no events were reported at the time of analysis for OS.

7. Secondary Outcome: Adverse Events
Description: All undesirable medical events experienced by the subject treated with the investigational product (including abnormal changes in laboratory values) are treated as adverse events and evaluated for safety.
Time Frame: Up to 30 months
Measure: Number; unit: participants
Arm/Group | SyB L-0501
Number analyzed (Participants) | 10
participants
  Any adverse event | 10
  Adverse drug reaction | 10
  SAE | 3
  Death | 0
  Discontinuation due to adverse events | 1
  Dose reduction due to adverse events | 5

8. Secondary Outcome: Number of Subjects With Clinically Significant Laboratory Test Values of Grade 3 or More
Description: Abnormalities in laboratory test values in overall study period were analyzed. Severity of abnormalities were evaluated using Common Terminology Criteria for Adverse Events (CTCAE). grade 1 : mild grade 2 : moderate grade 3 : severe or medically significant but not immediately life-threatening grade 4 : life threatening or disabling grade 5 : death related to adverse event
Time Frame: Up to 30 months
Measure: Number; unit: participants
Arm/Group | SyB L-0501
Number analyzed (Participants) | 10
participants
  CD4 lymphocytes decreased | 8
  Hyperglycemia | 1
  White blood cell decreased | 7
  Lymphocyte count decreased | 9
  Neutrophil count decreased | 8
  Platelet count decreased | 2

9. Secondary Outcome: Number of Subjects With Clinically Significant Physical Examination Values
Description: Number of subjects with abnormal or severe values of vital signs, electrocardiogram, and physical examination including ECOG performance status
Time Frame: Up to 30 months
Measure: Number; unit: participants
Arm/Group | SyB L-0501
Number analyzed (Participants) | 10
participants
  Vital signs | 0
  Electrocardiogram | 0
  Physical examination | 0

ADVERSE EVENTS:
Arm/Group | SyB L-0501
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SyB L-0501 (N=10)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1)
Ilium fracture (Injury, poisoning and procedural complications) | 1 (1)
Cytomegaloviral infection (Infections and infestations) | 1 (1)
Adenocarcinoma gastric (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SyB L-0501 (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (8)
Xerostomia (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (8)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Allergic colitis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Malaise (General disorders) | 5 (5)
Oedema peripheral (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Hypogammaglobulinemia (Immune system disorders) | 1 (1)
Conjunctivitis (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1)
Oral candidosis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Pain caused by treatment (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 4 (4)
Blood albumin decreased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Blood immunogloblin A decreased (Investigations) | 3 (3)
Blood immunogloblin G decreased (Investigations) | 3 (3)
Blood immunogloblin M decreased (Investigations) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Blood urea increased (Investigations) | 1 (1)
Blood uric acid decreased (Investigations) | 2 (2)
CD4 lymphocytes decreased (Investigations) | 10 (10)
Electrocardiogram QT prolonged (Investigations) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (2)
Hematocrit decreased (Investigations) | 2 (2)
Haemoglobin decreased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 9 (9)
Neutrophil count decreased (Investigations) | 10 (10)
Neutrophil count increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 9 (9)
Red blood cell count decreased (Investigations) | 2 (2)
Reticulocyte decreased (Investigations) | 2 (2)
Weight decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 9 (9)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Positional vertigo (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acneform dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Maculopapular rash (Skin and subcutaneous tissue disorders) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Phlebitis (Vascular disorders) | 2 (2)
Angialgia (Vascular disorders) | 2 (2)
Angiitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No